CLINICAL TRIAL: NCT04015635
Title: A Study of the Roles of the Immune and Inflammatory Systems in Hypertension
Brief Title: The Role of the Immune and Inflammatory Systems in Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Collaborators: European Research Council (Other)
Responsible Party: Principal Investigator, TOMASZ GUZIK, Prinicipal Investigator; Professor, University of Glasgow
Other Study IDs: 300798-01
Record Dates: First submitted 2019-04-30; First posted 2019-07-11 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Hypertension; Inflammation; Vascular Diseases
Keywords: blood pressure; hypertension; inflammation; immune dysfunction; endothelial dysfunction
MeSH Terms: conditions — Hypertension; Inflammation; Vascular Diseases; Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for flow cytometry. Blood and urine for biomarker analysis. Blood for possible RNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: 80 with hypertension, defined on office BP readings and confirmed with ambulatory blood pressure monitoring.
  Clinical and laboratory assessment. NO intervention.
  Interventions: Other: None involved
- Control: 80 WITHOUT hypertension, defined on office BP readings and confirmed with ambulatory blood pressure monitoring.
  Clinical and laboratory assessment. NO intervention.
  Interventions: Other: None involved

INTERVENTIONS:
Other: None involved — NO intervention

SUMMARY:
To define the cytokine and cellular immune signature of primary hypertension. Cross sectional clinical/laboratory study.

DETAILED DESCRIPTION:
Experimental data show the presence of immune and inflammatory systems dysregulation in hypertension. Understanding of the inflammatory and immune nature of hypertension is currently based on studies in rodent models of hypertension, but is supported by human epidemiological and genome wide association studies (GWAS) studies. It is now essential to identify key checkpoints and inflammatory mechanism(s) involved in human hypertension in comprehensive and sufficiently powered studies, which will then be able to guide subsequent in-depth hypothesis-driven mechanistic studies. This approach may provide the basis for future randomized clinical trials (RCTs).

To define the relationships and predictive value of the immune signature of hypertension and clinical phenotypes of hypertension :

* Predictive value of immune signature for blood pressure parameters measured by ambulatory blood pressure measurements (ABPM)
* Predictive value of immune signature for endothelial function assessed by Endo-PAT2000 and flow mediated dilatation (FMD) both complementary non-invasive techniques.
* Predictive value of immune signature for vascular stiffness and central pressure assessed by SphygmoCor
* Predictive value of immune signature for renal function parameters
* Predictive value of immune signature for cognitive function. To define genetic determinants of immune signature of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-55 years
* Cases: Office blood pressure ≥140 and ≥90
* Controls: Office blood pressure <140 and <90 and age, sex and BMI matching to cases

Exclusion Criteria:

* Age >55 years old;
* Secondary hypertension (including e.g. adrenal tumours, pheochromocytoma, renal artery stenosis; thyroid disease)
* Acute inflammatory disorders incl. flu, rhinitis, sinusitis etc. within 3 weeks;
* hospitalization within the past 3 months;
* Life expectancy of < 3 years;
* History of alcohol/substance abuse
* Inflammatory conditions e.g. Allergic disorders; chronic infections, COPD, tuberculosis; hepatitis B or C; pneumonitis, bronchiectasis; pericardial or pleural effusion, ascites; liver disease;
* Chronic inflammatory/autoimmune conditions such (e.g. SLE, rheumatoid arthritis, ulcerative colitis/Crohn's disease; non-basal cell malignancy or myelo- or lymphoproliferative disease within the past 5 years; known HIV+; Immunizations (3 months); pulmonary hypertension;
* Pregnancy, nursing;
* History of symptomatic coronary artery disease (events) or heart failure;
* BMI>40,
* diabetes/glucose intolerance (fasting glucose, HbA1; testing, glucose challenge where indicated);
* Known albuminuria/microalbuminuria;
* GFR<60mL/min/1.73m2.
* Any chronic concurrent treatment: Use of systemic or local steroids/immunosuppressive agents (within 6 months) of the inclusion; Current (within past 3 months) use of anti-hypertensive medication;
* Major depressive illness or other psychiatric conditions.
* Participants who decline participation in the study or who are unable to provide informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Otherwise fit and healthy individuals with hypertension who are treatment naive.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
cellular immune signature of primary hypertension: flow cytometry quantification of peripheral blood monocyte subtypes | rolling analysis until total number recruited or end of study period (June 2021)
  measuring expression of B cells markers, T cell markers, and DC cell markers
demographics: blood pressure | rolling analysis until total number recruited or end of study period (June 2021)
  systolic and diastolic; office and ambulatory; in mmHG
demographics: BMI | rolling analysis until total number recruited or end of study period (June 2021)
  in kg/m^2; calculated from height in meters and weight in kg

SECONDARY OUTCOMES:
Endo-PAT2000 "hyperaemia index" | until total number recruited or end of study period (June 2021)
  As a measure of endothelial function: measuring Peripheral Arterial Tone (PAT) signal changes to a reactive hyperemia challenge. The PAT signal is a measure of the digital pulsatile volume. The expected response is of a post occlusion increase of the PAT signal amplitude. PAT score is provided automatically by the system's software and is basically the ratio between the post- to pre- occlusion average signal size, corrected for systemic changes and baseline level.
  changes
flow mediated dilatation (FMD) (percent) | until total number recruited or end of study period (June 2021)
  as a measure of endothelial function
carotid intimal media thickness (mm) | until total number recruited or end of study period (June 2021)
  measure of vascular stiffness and central pressure
assessed by SphygmoCor (meters/second) | until total number recruited or end of study period (June 2021)
  measure of vascular stiffness and central pressure
serum Creatinine (mMol/L) | until total number recruited or end of study period (June 2021)
  measure of renal function
"International Physical Activity Questionnaire" (score) | until end of study period (June 2021)
  Questionnaire measures of physical activity. From hours of sedentary time, mild/moderate/vigorous activity over a week, it then calculates METs/week.
Interheart Diet Questionnaire score | until end of study period (June 2021)
  Questionnaire measures of health and activity. Based on known risk factors ie smoking diabetes, family history, dietary factors. Used as a validated measure of cardiovascular risk; score from 0 (minimal risk) to 48 (high risk)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Facility, Glasgow, City of Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Murray EC, Delles C, Orzechowski P, Renc P, Sitek A, Wagenaar J, Guzik TJ. Vascular phenotypes in early hypertension. J Hum Hypertens. 2023 Oct;37(10):898-906. doi: 10.1038/s41371-022-00794-7. Epub 2022 Dec 17. PMID 36528682

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT04015635/Prot_SAP_000.pdf